CLINICAL TRIAL: NCT05184634
Title: Determination of Physical Activity Levels,Quality of Life,Depression and Fatigue Severity of Individuals With Metabolic Syndrome
Brief Title: Determination Physical Activity Levels,Quality Life,Depression and Fatigue Severity Individuals With Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Büşra Sarıkaya (Other)
Responsible Party: Sponsor-Investigator, Büşra Sarıkaya, Physiotherapist, Kırıkkale University
Organization: Kırıkkale University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Screening
Other Study IDs: KÜ-BSarıkaya-001
Record Dates: First submitted 2021-12-06; First posted 2022-01-11 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome | interventions — Quality of Life

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Working group (Active Comparator): The data of the control group will be compared with the data of the study group.
  Interventions: Other: PHYSICAL ACTIVITY LEVELS; Other: DEPRESSION LEVELS; Other: FATİGUE SEVERİTY; Other: QUALITY OF LIFE
- Control Group (Active Comparator): The data of the study group will be compared with the data of the control group.
  Interventions: Other: PHYSICAL ACTIVITY LEVELS; Other: DEPRESSION LEVELS; Other: FATİGUE SEVERİTY; Other: QUALITY OF LIFE

INTERVENTIONS:
Other: PHYSICAL ACTIVITY LEVELS — Determination of physical activity levels of MetS individuals
Other: DEPRESSION LEVELS — To determine the depression levels of MetS individuals
Other: FATİGUE SEVERİTY — To determine the severity of fatigue of MetS individuals
Other: QUALITY OF LIFE — To determine the quality of life of MetS individuals

SUMMARY:
The aim of the study was to determine the Physical Activity Levels, Quality of Life, Depression and Fatigue Severity of Individuals with Metabolic Syndrome. International Physical Activity Questionnaire (IPAQ) to evaluate the physical activity level of individuals diagnosed with Metabolic Syndrome, to evaluate their quality of life SF-36 will be used to determine depression levels, Beck Depression Scale, and Fatigue Severity Scale (FSS) will be used to evaluate fatigue severity.

DETAILED DESCRIPTION:
Individuals who were diagnosed with metabolic syndrome and volunteered to participate in the study will be included in our study. The number of individuals was determined according to the power analysis. G*Power (version 3.1.9.4) package program was used for power analysis. As a result of the power analysis made assuming that the effect size that can be obtained between the two groups will be large (d= 0.451 (EFFECT YOU), at least 214 people were included in the study (at least 107 people for each group)) at a 95% confidence level (with a margin of error of 0.05). It was calculated that 95% power could be obtained.After determining the number of individuals, the same number of normal healthy individuals who were not diagnosed with metabolic syndrome will be included in the study as the control group.Scales will be used to determine physical activity levels, Quality of life, Depression and Fatigue Severity in the control and study groups. Physical activity The International Physical Activity Questionnaire (IPAQ) will be used to assess the level of life, SF-36 will be used to assess their quality of life, the Beck Depression Scale will be used to determine depression levels, and the Fatigue Severity Scale (FSS) will be used to assess the severity of fatigue.

Demographic information (name, surname, age, education level, occupation, marital status, background, family history, disease history, medication, smoking and alcohol use, regularly used drugs) of the individuals who will participate in the study will be recorded in the patient evaluation form.

The International Physical Activity Questionnaire (IPAQ) will be used to assess the level of physical activity, the SF-36 will be used to assess their quality of life, the Beck Depression Scale will be used to determine depression levels, and the Fatigue Severity Scale (FSS) will be used to assess the severity of fatigue.

International Physical Activity Questionnaire (IPAQ): Physical activity level will be assessed with the short version of the IPAQ. The walking duration of the individuals in the last 1 week will be determined in terms of MET-minutes/week, whether they did moderate and severe PA, and if they did, how many days per week and total minutes they did. As a result, all values are added together to determine the total IPAQ score and will be categorized as inactive, minimally active, and very active.

Quality of Life Scale-Short Form (SF-36) Form: It was collected with Quality of Life Scale-Short Form (SF 36). The Quality of Life Scale is accepted and applied as an individual's quality of life assessment scale. SF-36 was developed by Hays, Wells, Sherbourne, Rogers, and Spritzer (1995), and its Turkish reliability and validity study was performed by Koçyiğit, Aydemir, Ölmez, Fişek, and Memiş (1999). The SF-36 is a self-report scale and examines eight dimensions of health with 36 items, such as physical functioning, social functioning, role difficulties (physical and emotional), mental health, vitality (vitality), pain, and general perception of health. The scale provides an evaluation between zero and 100, and a higher score indicates a better level of health.

Beck Depression Inventory (BDI): It is a self-assessment scale applied to healthy and psychiatric patient groups. Its purpose is to determine the risk for depression and to measure the level and severity of depressive symptoms. This form, which includes a total of 21 self-evaluation scales, provides a four-point Likert type measurement. Each item gets an increasing score between 0-3 and the total score is obtained by summing them up. A high total score indicates a high level of depression severity. It was developed by Beck et al. and adaptation, validity and reliability studies were conducted for the Turkish population. In the Turkish validity and reliability article of the scale, the cut-off point was determined as 17.

Fatigue Severity Scale (FAS): In the evaluation of the fatigue levels of the individuals, the Turkish validity and reliability of the TLS was used. This scale consists of nine items. Each item is scored between 1 and 7, and as the total score decreases, so does fatigue.

The data will be analyzed with the SPSS package program. Appropriate statistical analysis will be made.

After the data are obtained, it is aimed to evaluate the results and write a scientific thesis and publish it in an international journal.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of metabolic syndrome
* to work as a volunteer those who agreed to participate

Exclusion Criteria:

* No surgery in the last 3 months
* with communication problem

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2021-12-15 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-07-04 (Actual)

PRIMARY OUTCOMES:
Physical Activity Levels | 3 minute
  International Physical Activity Questionnaire (IPAQ): Physical activity level will be assessed with the short version of the IPAQ. The walking duration of the individuals in the last 1 week will be determined in terms of MET-minutes/week, whether they did moderate and severe PA, and if they did, how many days per week and total minutes they did. As a result, all values are added together to determine the total IPAQ score and will be categorized as inactive, minimally active, and very active.
Life quality | 3 minute
  Quality of Life Scale-Short Form (SF-36) Form: It was collected with Quality of Life Scale-Short Form (SF 36). The Quality of Life Scale is accepted and applied as an individual's quality of life assessment scale. SF-36 was developed by Hays, Wells, Sherbourne, Rogers, and Spritzer (1995), and its Turkish reliability and validity study was performed by Koçyiğit, Aydemir, Ölmez, Fişek, and Memiş (1999). The SF-36 is a self-report scale and examines eight dimensions of health with 36 items, such as physical functioning, social functioning, role difficulties (physical and emotional), mental health, vitality (vitality), pain, and general perception of health. The scale provides an evaluation between zero and 100, and a higher score indicates a better level of health.
Depression Levels | 3 minute
  Beck Depression Inventory (BDI): It is a self-assessment scale applied to healthy and psychiatric patient groups. Its purpose is to determine the risk for depression and to measure the level and severity of depressive symptoms. This form, which includes a total of 21 self-evaluation scales, provides a four-point Likert type measurement. Each item gets an increasing score between 0-3 and the total score is obtained by summing them up. A high total score indicates a high level of depression severity. It was developed by Beck et al. and adaptation, validity and reliability studies were conducted for the Turkish population. In the Turkish validity and reliability article of the scale, the cut-off point was determined as 17.
Fatigue Severity | 3 minute
  Fatigue Severity Scale (FAS): In the evaluation of the fatigue levels of the individuals, the Turkish validity and reliability of the TLS was used. This scale consists of nine items. Each item is scored between 1 and 7, and as the total score decreases, so does fatigue.

CONTACTS AND LOCATIONS:
Locations (1):
- Kırıkkale Üniversitesi, Kırıkkale, Turkey (Türkiye)